CLINICAL TRIAL: NCT02681562
Title: A Phase II, Open Label, Controlled Study of Olaparib in Locally Advanced ER, PgR and HER2 Negative (Triple Negative) and in Locally Advanced Germline BRCA Mutation-positive Breast Cancer Patients: Biological Evaluation From a "Window of Opportunity" Trial
Brief Title: Olaparib in Locally Advanced ER, PgR and HER2 Negative (Triple Negative) and in Locally Advanced Germline BRCA Mutation-positive Breast Cancer Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Istituti Ospitalieri di Cremona (Other)
Responsible Party: Principal Investigator, Giandomenico Roviello, Medical Doctor, Istituti Ospitalieri di Cremona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ISS22810078
Record Dates: First submitted 2016-02-08; First posted 2016-02-12 (Estimated); Last update posted 2016-02-15 (Estimated); Status verified 2016-02

CONDITIONS: Breast Cancer; Triple Negative Breast Cancer
Keywords: olaparib
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — olaparib

ARMS (2):
- Olaparib triple negative (Experimental): Olaparib short administration in triple negative breast cancer
  Interventions: Drug: olaparib
- Olaparib BRCA mutated (Experimental): Olaparib short administration in BRCA mutated patients
  Interventions: Drug: olaparib

INTERVENTIONS:
Drug: olaparib

SUMMARY:
Treatment selection for breast cancer is still largely empiric and guided by large randomized clinical trials on populations of patients. This approach is inadequate for the selection of individualized chemotherapy regimens. Estimates of benefits for individuals are extrapolations from the effects seen in these large trials, and do not necessarily apply to individual patients. The revolution in genomics promises to transform oncology care. By better defining cancer subtypes, a better understanding of breast cancer biology should help to guide treatment.

The up-front phase we have decide to adopt play a pivotal role as it is useful for testing a targeted therapeutic drug such as olaparib wich also requires development of new biomarkers which may be useful for future studies. With this approach it could be possible to demonstrate drug target or biomarker effect in clinical setting and models the relationship between the pharmacodynamics and the pharmacokinetics. Additional benefits of this approach include the following:

* It could facilitate rational drug selection, identify therapeutic failures early, and compress timelines for anticancer drug development.
* It could provide initial rationale and guiding principles for further drug development based on studies in humans (rather than xenografts, where tissues of one species are transplanted to another species).
* As it focuses on extensively characterizing how a drug works and whether it hits its intended target (including molecular imaging studies) in a limited number of patients it could yield results that would optimally inform and expedite the subsequent development of molecularly-targeted agents

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study specific procedures
2. Patients (female) must be 18 years of age.
3. Clinically or radiologically measurable or evaluable disease defined as: presence of bidimensionally or unidimensionally measurable breast lesion by physical or radiological examination.
4. Estrogen receptor < 10% for ARM A only
5. Progesterone receptor = 0 for ARM A only
6. HER2 negative on primary tumor (HER-2 score of 0 or 1+/2+ with FISH not amplified) for ARM A only
7. Mutation of BRCA 1 and/or 2 for ARM B only

   * Germline BRCA1 or BRCA2 mutation that is considered deleterious or suspected deleterious (include those mutations or translocations termed "deleterious" or "suspected deleterious" according to lab reporting). Testing under the context of this protocol may be performed at any time prior to allocation.
   * Patients who have a prior BRCA test may be enrolled into the study based at the result of the prior test
   * Provision of informed consent for genetic research. If a patient declines to participate in the genetic research, there will be no penalty or loss of benefit to the patient. The patient will not be excluded from other aspects of the study described in this Clinical Study Protocol, so long as they consent to that part.
8. Patients must have normal organ and bone marrow function, ECOG performance status 0-1 (can be amended for specific populations studies)
9. Adequate cardiac function: left ventricular ejection fraction (LVEF) at rest measured by echocardiography must be no lower than the local normal limit.
10. Absence of clinically significant cardiovascular disease (e.g. myocardial infarction, unstable angina), New York Hearth Association (NYHA) grade II or greater congestive hearth failure, serious cardiac arrhythmia requiring medication, or grade II or greater peripheral vascular disease within 12 months prior to day 1 on study
11. Patients must have voluntarily agreed to participate by given informed consent. Written informed consent must be dated and signed by both patients and investigator

Exclusion Criteria:

1. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site)
2. Previous enrolment in the present study
3. Participation in another clinical study with an investigational product during the last 12 months
4. Any previous treatment with a PARP inhibitor, including olaparib.
5. Patients receiving any systemic chemotherapy, radiotherapy (except for palliative reasons), within 2 weeks from the last dose prior to study treatment (or a longer period depending on the defined characteristics of the agents used). The patient can receive a stable dose of bisphosphonates for bone metastases, before and during the study as long as these were started at least 4 weeks prior to treatment with study drug.
6. Concomitant use of known CYP3A4 inhibitors such as ketokonazole, itraconazole, ritonavir, indinavir, saquinavir, telithromycin, clarithromycin and nelfinavir
7. Blood transfusions within 1 month prior to study start
8. Patients with myelodysplastic syndrome/acute myeloid leukaemia.
9. Patients with-out any sign or symptoms of distant metastases.
10. Major surgery within 14 days of starting study treatment and patients must have recovered from any effects of any major surgery.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2016-01; Primary Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between baseline gene and protein expression profile and clinical response | Duration of the study

SECONDARY OUTCOMES:
Assess overall response rate by RECIST criteria evaluated clinically in each treatment group | Through study completion, an average of 1 year
Evaluate safety and tolerability of olaparib alone assessed by CTCAE v4.0 | Through study completion, an average of 1 year
Compare time to deterioration of health-related quality of life by QLQ-C30 scale | Through study completion, an average of 1 year
Compare health status by QLQ-C30 scale | Through study completion, an average of 1 year

REFERENCES:
- [Derived] Roviello G, Milani M, Gobbi A, Dester M, Cappelletti MR, Allevi G, Aguggini S, Ravelli A, Gussago F, Cocconi A, Zanotti L, Senti C, Strina C, Bottini A, Generali D. A Phase II study of olaparib in breast cancer patients: biological evaluation from a 'window of opportunity' trial. Future Oncol. 2016 Oct;12(19):2189-93. doi: 10.2217/fon-2016-0116. Epub 2016 Jun 21. PMID 27324108